CLINICAL TRIAL: NCT03649529
Title: Adoptive Immunotherapy for HLA_A2 Genotype gp100 Positive Malignant Melanoma With GPA-TriMAR-T Cell
Brief Title: Treatment of Malignant Melanoma With GPA-TriMAR-T Cell Therapy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Collaborators: The Second Affiliated Hospital of Hainan Medical University (Other); Hainan Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T2018-7
Record Dates: First submitted 2018-08-23; First posted 2018-08-28 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Malignant Melanoma
Keywords: HLA-A2; gp100
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Patients' autologous T cells will be isolated and transduced by GPA-TriMAR lentivirus to generate the GPA-TriMAR-T cells,and then infused back into the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GPA-TriMAR-T (Experimental): Patients' autologous T cells will be isolated and transduced by GPA-TriMAR lentivirus to generate the GPA-TriMAR-T cells, and these cells will then be infused back into the patient for intervention.
  Interventions: Biological: GPA-TriMAR-T

INTERVENTIONS:
Biological: GPA-TriMAR-T — Patients will undergo leukapheresis to isolate autologous T cells, these T cells will be activated and modified to express GPA-TriMAR in the manufacture facility, and eventually infused back into the body for treatment.
  Other Names: TCR-mimic-CAR-T

SUMMARY:
Malignant melanoma have been reported to be characterized with high gp100 expression. Patients' autologous T cells will be isolated and transduced by GPA-TriMAR lentivirus to generate the GPA-TriMAR-T cells. When infused back to the patient, the GPA-TriMAR-T cells will recognize and kill target cells that express gp100(209-217) peptides in the form MHC-I complex, thus eliminating malignant melanoma from the body.

DETAILED DESCRIPTION:
GPA-TriMAR is a modified chimeric antigen receptor (CAR) that consist of three subunit in it's outer membrane domain. The outer membrane domain linked to the inner membrane 4-1BB/CD3ζ domain through the transmembrane domain, thus compose the complete chimeric antigen receptor. Patients' autologous T cells will be isolated and transduced by GPA-TriMAR lentivirus to generate the GPA-TriMAR-T cells. When infused back to the patient, the modified GPA-TriMAR-T cells will recognize and kill malignant melanoma cells in the body, and in the meanwhile the other two subunits function to stimulate the innate immune system and enhance GPA-TriMAR-T cells tumor Infiltration.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must personally sign and date the consent form before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. HLA_A2 genotype and gp100 positive malignant melanoma： Ⅳ stage or relapsed after surgery or chemotherapy or no available standard therapy;
4. At least one measurable lesion per RECIST V1.1;
5. Aged 18 to 69 years;
6. Expected survival ≥12 weeks; Eastern cooperative oncology group (ECOG) performance status of≤2;
7. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
8. All other treatment induced adverse events must have been resolved to ≤grade 1;
9. Laboratory tests must fulfill the following criteria: ANC ≥ 1000/uL, HGB>70g/L, Platelet count ≥ 50,000/uL, Creatinine clearance ≤1.5 ULN, Serum ALT/AST ≤2.5 ULN, Total bilirubin ≤1.5 ULN (except in subjects with Gilbert's syndrome);

Exclusion Criteria:

1. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring iv antimicrobials for management. (Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment);
2. Patients with symptomatic central nervous system metastasis, intracranial metastasis, and cancer cells found in cerebrospinal fluid are not recommended to participate in this study. Symptom free or post-treatment stable disease or disappearance of lesions should not be excluded. The specific selection is ultimately determined by the investigator;
3. Lactating women or women of childbearing age who plan to conceive during the time period;
4. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
5. Known history of infection with HIV;
6. Subjects need systematic usage of corticosteroid;
7. Subjects need systematic usage of immunosuppressive drug;
8. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
9. Other reasons the investigator consider the patient may not be suitable for the study.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-09-27 (Actual); Primary Completion 2021-09-15 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
safety （Incidence of treatment-related adverse events as assessed by CTCAE v4.03） | 24 months
  Incidence of treatment-related adverse events as assessed by CTCAE v4.03

SECONDARY OUTCOMES:
Complete response rate[CR] （Complete response rate per the revised International Working Group (IWG) Response Criteria） | 24 months
  Complete response rate per the revised International Working Group (IWG) Response Criteria
Partial response rate [PR] （Partial response rate per the revised International Working Group (IWG) Response Criteria） | 24 months
  Partial response rate per the revised International Working Group (IWG) Response Criteria
Duration of Response （The time from response to relapse or progression） | 24 months
  The time from response to relapse or progression
Progression Free Survival （The time from the first day of treatment to the date on which disease progresses.） | 24 months
  The time from the first day of treatment to the date on which disease progresses.
Overall Survival （The number of patient alive, with or without signs of cancer） | 24 months
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Lin, Principal Investigator — The Second Affiliated Hospital of Hainan Medical University
Locations (2):
- China (2):
  - Hainan Cancer Hospital, Haikou, Hainan
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang G, Wang L, Cui H, Wang X, Zhang G, Ma J, Han H, He W, Wang W, Zhao Y, Liu C, Sun M, Gao B. Anti-melanoma activity of T cells redirected with a TCR-like chimeric antigen receptor. Sci Rep. 2014 Jan 6;4:3571. doi: 10.1038/srep03571. PMID 24389689
- [Background] Zhang G, Liu R, Zhu X, Wang L, Ma J, Han H, Wang X, Zhang G, He W, Wang W, Liu C, Li S, Sun M, Gao B. Retargeting NK-92 for anti-melanoma activity by a TCR-like single-domain antibody. Immunol Cell Biol. 2013 Nov-Dec;91(10):615-24. doi: 10.1038/icb.2013.45. Epub 2013 Oct 8. PMID 24100387
- [Background] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994